CLINICAL TRIAL: NCT06821152
Title: A Functional Performance and Acceptability Evaluation of the Miss Liberty Female Condom Compared to the FC2 Female Condom
Brief Title: Functional Performance and Acceptability Evaluation of the Miss Liberty Female Condom Compared to the FC2 Female Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Prof Mags Beksinska, Executive Director, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Miss Liberty
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Functional Performance
Keywords: Female condom; condom acceptability; Miss Liberty; FC2; condom safety

STUDY DESIGN:
Intervention Model Description: This research study will be a two-period, cross-over randomized controlled trial to compare the functional performance, safety and acceptability of two female condom types.
Who Masked: Outcomes Assessor
Masking Description: The statistician preparing the randomization sequences and analyzing the data will remain masked while developing and testing the analysis programs and procedures and drafting the preliminary study report.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Type A - Type B (Active Comparator): A separate randomization process (implemented by an independent statistician) will allocate one of the two study condom types to the letters A and B which will be used to label individual packs of five condoms for distribution to study women and to record the condom type used in each study period.
  Interventions: Device: Miss Liberty Condom; Device: FC2 condom
- Arm 2 -Type B - Type A (Active Comparator): A separate randomization process (implemented by an independent statistician) will allocate one of the two study condom types to the letters A and B which will be used to label individual packs of five condoms for distribution to study women and to record the condom type used in each study period.
  Interventions: Device: Miss Liberty Condom; Device: FC2 condom

INTERVENTIONS:
Device: Miss Liberty Condom — The Miss Liberty female condom is manufactured by Zhejiang Rui Bo 001 High Polymer Co, Ltd. The condom is designed as a loose-fitting pouch that lines the vagina. It has two flexible rings. The sheath, are made of polyurethane. The outer ring remains outside the vagina and covers the external genitalia during intercourse. An internal ring is removable and serves as the insertion mechanism and anchors the device within the vagina. Miss Liberty measures 180mm in length and 78mm in lay-flat width. The device is pre-lubricated with silicone oil. This condom is a similar design (material, length, width) to the USFDA approved FC1 female condom which was discontinued and replaced by FC2.
Device: FC2 condom — The FC2 is a second-generation female condom manufactured by the Female Health Company (Chicago, IL). The FC2 has US FDA approval and has been granted the CE Mark of the European Union. The FC2 is pre-qualified by the WHO. The condom is designed as a loose-fitting pouch that lines the vagina. It has two flexible rings. The outer ring at the open end is rolled from the nitrile material. The outer ring remains outside the vagina and covers the external genitalia during intercourse. An internal ring is removable and serves as the insertion mechanism and anchors the device within the vagina. FC2 measures 170mm in length and 80mm in lay-flat width. The device is pre-lubricated with silicone oil. This FC is available in the public health sector in South Africa.

SUMMARY:
The purpose of the study is to evaluate the functional performance and acceptability of the Miss Liberty female condom version 1 (Miss Liberty female condom), compared to the FC2 female condom.

The study will be a sequential randomised 2-period cross-over trial comparing five uses of the Miss Liberty female condom, compared to the control FC2 female condom. Each woman will be asked to use five Miss Liberty female condoms, and five FC2 control female condoms in a randomised order. Woman will complete a Condom Use Report after each condom use. Function, safety, and acceptability will be assessed at each of two follow-up visits conducted after using each set of five condoms. The trial will enrol 235 women between 18-45 years old.

The primary objective is to ascertain the functional performance of the Miss Liberty female condom compared to the control FC2 female condom. The secondary objectives are to determine the acceptability and safety (as determined by the number of adverse events) for the Miss Liberty female condom compared to the FC2 female condom.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the functional performance and acceptability of the Miss Liberty female condom version 1 (Miss Liberty female condom), compared to the FC2 female condom.

This research study will be a two-period, cross-over randomized controlled trial to compare the functional performance, safety and acceptability of two female condom types. Enrolled women will be asked to use five FC2, or five Miss Liberty female condoms in each study period provided to them in random order according to one of two possible sequences of each condom type. A Condom Use report will be completed after each condom use and a Condom Acceptability Questionnaire will be completed at the end of each study period after use of each set of five study condoms.

If a woman expresses interest in participating, she will be given the study information sheet to read, which will describe the study requirements including her role in the study. If she agrees to take part in the research, she will be invited to the Wits MRU Commercial City site and asked to provide written informed consent.

A physical examination will be undertaken to exclude visible symptoms of sexually transmitted infection. If symptoms are observed the participant will be referred to a Department of Health clinic or their doctor for treatment. A urine pregnancy test will be conducted at screening to exclude pregnancy. Woman will need to provide a copy of HIV testing results which are not older than two months. If HIV testing results are not available, voluntary HIV counselling and testing will be offered and conducted by study staff. Woman will be counselled on Pre Exposure Prophylaxis (PrEP) and referred to a local facility that provides PrEP should they wish to initiate PrEP.

The consent process and all checklists, condom use reports and questionnaires used in the research will be written and conducted in a language that is understandable to the participant, and all relevant documents will be translated into isiZulu.

Woman will be instructed on proper condom use. After successful completion of the screening process and documentation of informed consent the woman will be formally enrolled in the study and assigned the next consecutive participant Identification Number (PID). The Baseline Questionnaire covering information on participant demographics and previous female and male condom use will be administered in private. The study staff will discuss with the woman an approximate timeframe for use of all five condoms and a suitable follow-up date will be scheduled. This date will be noted on an appointment slip. Woman will be encouraged to come back if their condoms are finished before the due date and will be given the research study contact details to call for any appointment changes.

After successful completion of the screening process and documentation of informed consent the woman will be formally enrolled in the study and assigned the next consecutive PID.

Participants will be asked to return for a follow-up visit after using each set of five study condoms. There will be two follow-up visits. At each of these visits study staff will review the information on the condom reports for completeness and accuracy. Data on device function and safety (individual Condom Use Reports) for each condom type will be collected during follow-up visits.

Condom use instructions will be reviewed as a reminder before use of the next set of study condoms. The participation period for each study woman is expected to last between 2-3 months.

During the 1st in-person follow-up visit, women will be interviewed about their first assigned condom type and they will receive their next condom packet within their second randomly assigned use sequence. In the second follow-up visit, woman will be interviewed about their second assigned condom type and will be discontinued from study participation. If the woman experiences any failure event during sexual intercourse they will be offered HIV testing and STI testing (Chlamydia/gonorrhoea). Woman will be instructed to return any unopened condoms at the next visit. If a woman does not keep their scheduled follow-up visit, research personnel will initiate a reminder contact and reschedule the visit.

Each follow-up interview should be scheduled approximately one month after the preceding visit.

At the second follow-up visit, woman will return their five completed Condom Use Reports for the second set of condoms. Any missing or unclear responses on the Condom Use Reports will be clarified at this time. A Condom Acceptability Questionnaire will be completed at the visit. Woman who fail to return to the site for the second follow-up visit will be contacted by research staff to reschedule the visit.

Woman may discontinue from the study before the scheduled end. A woman which does not complete both study periods will be classified as an early discontinuer and classified as follows:

* Medical/safety reason(e.g. the female partner becomes pregnant, or has a sensitivity/allergic reaction to the research study products, or is diagnosed with a new onset sexually transmitted infection, etc.);
* Non-safety reason related to use of the research study products (e.g. she dislikes the research study products and/or fails to follow protocol requirements that are felt to significantly alter study outcomes);
* Non-safety reasons NOT related to use of the research study products (e.g. desires pregnancy, moves, relationship with partner dissolved, does not wish to continue, etc.);
* Loss-to-follow-up if a participating woman has not returned to the clinic for their scheduled follow-up visit and all efforts to locate them have failed.
* Investigator decision The investigator decides to discontinue the woman from the study for a safety or other study related circumstance.

Two hundred and thirty five eligible women willing to participate in the study will be randomized to condom use order. To minimize a potential learning effects, women will be randomly assigned to the sequence of use of condom type. Use-order assignments will be computer generated using REDCap. Women will be randomly assigned in balanced blocks of size 2, 4 or 6 chosen at random to one of two possible condom use sequences:

1. Type A - Type B
2. Type B - Type A

A separate randomization process (implemented by an independent statistician) will allocate one of the two study condom types to the letters A and B which will be used to label individual packs of five condoms for distribution to study women and to record the condom type used in each study period. Study staff will be masked to the extent possible until all data have been captured and the primary analysis programs have been verified. Due to physical differences between the study products (color, texture, width) masking study participants and clinic staff can only be assured during enrolment and collection of baseline data, but cannot be maintained throughout the study.

The statistician preparing the randomization sequences and analyzing the data will remain masked while developing and testing the analysis programs and procedures and drafting the preliminary study report. The date the statistician is unmasked will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 45 years (inclusive);
* Be of female sex and gender
* Be literate (able to read a newspaper or letter easily);
* Have been in an exclusive (monogamous) heterosexual sexual relationship with a male partner partner for at least 3 months; and intend to continue to be an exclusive (monogamous) sexual relationship with their spouse or partner while participating in this research study;
* Be sexually active (defined as having at least one vaginal coital act per week);
* Willing to give informed consent;
* Willing to complete the female condom coital use reports;
* Willing to use the study condoms as directed;
* Agree to only use the study condoms sequentially during time of participation
* Willing to adhere to the follow-up schedule and all study procedures;
* Willing to provide research study staff with an address, phone number or other locator information while participating in the study;
* Willing to participate in the study for the duration of 10 condom uses (approximately 2- 3 months);
* Willing to have a fingerprint scan to exclude co-enrolment in other research projects;
* Using hormonal or other non-barrier contraception (e.g. Oral Contraceptives, injectables, implant, Intrauterine device (IUD), or have had a tubal sterilization) or male partner vasectomised;
* Agree to return any unopened condoms;
* Agree to not bring study condoms in contact with genital or oral piercing jewelry;
* Able to understand instructions for correct use of female condoms;
* Agree not to use male condoms when using the female condom in a single sex act.

Exclusion Criteria:

* Woman is pregnant or desires to become pregnant during the time of the research study;
* Known to be HIV positive by self report;
* Self-reported history of current sexually transmitted infection (e.g. gonorrhea, syphilis, Chlamydia);
* Female (or reports her partner) has genital piercing jewelry, uses genital beading or uses sex toys, drugs, medications or non-study devices that can affect sexual performance;
* Female (or reports her partner) has known sensitivities or allergies to latex, synthetic nitrile, vaginal/sexual lubricants or lubricants used on condoms;
* Female has symptoms of a sexually transmitted infection (STI).
* Male partner has known erectile or ejaculatory dysfunction;
* Is a past or current employee of the University of the Witwatersrand or Miss Liberty Ltd;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be female as female condoms inserted vaginally are being evaluated
Enrollment: 235 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Clinical breakage | 2-3 months
  Defined as breakage or tearing of the female condom during sexual intercourse or during withdrawal from the vagina. Clinical breakage is breakage with potential adverse clinical consequences. The clinical breakage rate is calculated by dividing the number of female condoms reported to have broken or torn during sexual intercourse or during withdrawal by the number of female condoms used during sexual intercourse.
Clinical slippage | 2-3 months
  Defined as an instance when a female condom slips completely out of the vagina during sexual intercourse. The clinical slippage rate is calculated by dividing the number of female condoms that slipped by the number of female condoms used during sexual intercourse.
Clinical misdirection | 2-3 months
  Defined as vaginal penetration whereby the penis is inserted between the female condom and the vaginal wall. The clinical misdirection rate is calculated by dividing the number of reported events of misdirection by the number of female condoms used during sexual intercourse.
Clinical invagination | 2-3 months
  Defined as an instance when the external retention feature of the female condom is partially or fully pushed into the vagina during sexual intercourse.
  The clinical invagination rate is calculated by dividing the number of events of invagination by the number of female condoms used during sexual intercourse.
Total clinical failure | 2-3 months
  Defined as the sum of female condoms with at least one clinical failure event (clinical breakage, clinical slippage, clinical misdirection, clinical invagination) clinically break or additional failure modes(s) identified in the risk assessment which results in the reduction of the female condom protective function. The total clinical failure rate is calculated by dividing the number of female condoms with a clinical failure by the number of female condoms used during sexual intercourse.

SECONDARY OUTCOMES:
Condom Safety | 2-3 months
  Rates of genital discomfort reported to have occurred during or immediately after condom use. Genital adverse events will be classified by relatedness, expectedness and severity
Acceptability | 2-3 months
  Frequency of key acceptability outcome measures will be calculated and include: comfort in use; ease of insertion and removal; like or dislike of product attributes; adequacy and feel of lubrication and sensitivity and stimulation.
Non-Clinical breakage | 2-3 months
  Defined as breakage noticed before sexual intercourse or occurring after withdrawal of the female condom from the vagina. Non-clinical breakage is breakage with no potential adverse clinical consequences. The non-clinical breakage rate is calculated by dividing the number of female condoms reported to have broken before sexual intercourse or after withdrawal by the number of female condom packages opened
Total breakage | 2-3 months
  Defined as the sum of all female condom breakages at any time before, during or after sexual intercourse. It includes both clinical breakages and non-clinical breakages. The total breakage rate is calculated by dividing the total number of female condoms that broke by the number of female condom packages opened.
Non-Clinical slippage | 2-3 months
  Defined as slippage when the female condom slips/ moves out of the vagina but not completely. Non-clinical slippage is slippage with no potential adverse clinical consequences. The non-clinical slippage rate is calculated by dividing the number of female condoms reported to have partially slipped during sexual intercourse by the number of female condoms used during vaginal intercourse

CONTACTS AND LOCATIONS:
Overall Officials: Mags Beksinska, PhD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- MatCH Research Unit [Maternal, Adolescent and Child Health Research Unit], Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holm S. A simple sequentially rejective multiple test procedure. Scand J Statist 6: 65-70, 1979).
- [Background] Taylor D. Issues in the design, analysis and interpretation of condom functionality studies. Contraception. 2009 Sep;80(3):237-44. doi: 10.1016/j.contraception.2009.03.004. Epub 2009 Apr 23. PMID 19698815
- [Background] Beksinska M, Wong R, Smit J. Male and female condoms: Their key role in pregnancy and STI/HIV prevention. Best Pract Res Clin Obstet Gynaecol. 2020 Jul;66:55-67. doi: 10.1016/j.bpobgyn.2019.12.001. Epub 2019 Dec 14. PMID 32007451
- [Background] Center for Health and Gender Equity. Female condoms and US foreign assistance: an unfinished imperative for women's health. Washington, DC; 2011
- [Background] United Nations Population Fund. HIV prevention gains momentum. New York: UNFPA, 2011. 978-0-89714-933-4
- [Background] Shisana O, Rehle T, Simbayi LC, et al. South African national HIV prevalence, incidence, behaviour and communication survey 2017: Health and wellbeing: Human Science Research Council Press; 2017
- [Background] Martinez G, Copen CE, Abma JC. Teenagers in the United States: sexual activity, contraceptive use, and childbearing, 2006-2010 national survey of family growth. Vital Health Stat 23. 2011 Oct;(31):1-35. PMID 22256688
- [Background] Warren M. Condoms: the multipurpose prevention technologies that already exist. BJOG. 2014 Oct;121(Suppl 5):9-11. doi: 10.1111/1471-0528.12913. No abstract available. PMID 25335833
- [Background] World Health Organization Department of Sexual and Reproductive Health and Research (WHO/SRH) and Johns Hopkins Bloomberg School of Public Health/ Center for Communication Programs (CCP), Knowledge SUCCESS. Family Planning: A Global Handbook for Providers (2022 update). Baltimore and Geneva: CCP and WHO; 2022. chromeextension://efaidnbmnnnibpcajpcglclefindmkaj/https://fphandbook.org/sites/default/files/WH O-JHU-FPHandbook-2022Ed-v221114b.pdf
- See also: UNFPA, Universal access to Reproductive Health: Progress and Challenges. — https://www.unfpa.org/sites/default/files/pub-pdf/UNFPA_Reproductive_Paper_20160120_online.pdf
- See also: Muchiri E, Odimegwu E, DeWet N. HIV risk perception and consistency in condom use among adolescents and young adults in urban Cape Town, South Africa: a cumulative risk analysis. S Afr J Infect Dis [Internet]. 2017 [cited 2019 Sep 8]; 32(3):105-110. — https://doi.org/10.1080/23120053.2017.1332800
- See also: eproductive Health Supplies Coalition. Caucus on new and underused reproductive health technologies. Product brief: female condom. Reproductive Health Supplies Coalition; 2013. [Online]. [Cited: 19th Dec 2016]. — https://www.rhsupplies.org/uploads/tx_rhscpublications/RHSC_fem_condom_br.pdf
- See also: UNFPA Prequalified Female Condom Manufacturers List — https://www.unfpa.org/resources/unfpa-prequalified-female-condom-manufacturers-list
- See also: ISO 29943-2:2017 Condoms - Guidance on clinical studies - Part 2: Female condoms, clinical function studies based on self-diaries. — https://www.iso.org/standard/62497.html
- See also: ISO 25841:2017 Female condoms Requirements and test methods. — https://www.iso.org/standard/66676.html